CLINICAL TRIAL: NCT03470571
Title: Predictive Value of CMR Features in Patients With Suspected Myocarditis
Brief Title: CMR Features in Patients With Suspected Myocarditis
Acronym: CMRMyo
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Raymond Y. Kwong, MD, Associate Professor of Medicine, Harvard Medical School, Brigham and Women's Hospital
Other Study IDs: CMR Myocarditis
Record Dates: First submitted 2018-03-13; First posted 2018-03-20 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Outcome, Fatal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CMR — Outcome analysis of CMR features in suspected myocarditis patients

SUMMARY:
Presentation of myocarditis is heterogeneous, often ranges from being asymptomatic, to chest pain, dyspnoea, palpitations, and even sudden cardiac death. Diagnosing myocarditis is challenging with no current uniform clinical gold-standard. CMR is a key investigative tool, however the predictive value of CMR features is unknown. In this study we assess 670 consecutive patients with suspected myocarditis who were referred for CMR between 2002 and 2015 at the BWH. CMR features such as late gadolinium sizing, T1 mapping, extracellular volume fraction assessment, strain analysis (feature tracking), clinical data, labortory tetsings and electrocardiogramm are linked to the outcome in order to assess its predictive value.

ELIGIBILITY:
Inclusion Criteria:

* patients referred by their treating physician to undergo CMR for "suspected myocarditis" as the primary clinical question

Exclusion criteria

* evidence of coronary artery disease
* hypertrophic cardiomyopathy
* arrhythmogenic right ventricular cardiomyopathy
* cardiac sarcoidosis
* cardiac amyloidosis
* takotsubo cardiomyopathy
* constrictive pericarditis
* Loeffler endocarditis
* ventricular non-compaction
* cardiac tumor
* pulmonary embolism
* severe valve disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study includes consecutive patients referred by their treating physician to undergo CMR for "suspected myocarditis" as the primary clinical question between December 2002 and December 2015 at our center.
Sampling Method: Non-Probability Sample
Enrollment: 670 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac events | through study completion, an average of 2 years
  Heart failure hospitalization; all cause death; sustained ventricular arrhythmia; recurrent myocarditis; transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Shapiro Cardiovascular Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bernhard B, Tanner G, Garachemani D, Schnyder A, Fischer K, Huber AT, Safarkhanlo Y, Stark AW, Guensch DP, Schutze J, Greulich S, Bastiaansen JAM, Pavlicek-Bahlo M, Benz DC, Kwong RY, Grani C. Predictive value of cardiac magnetic resonance right ventricular longitudinal strain in patients with suspected myocarditis. J Cardiovasc Magn Reson. 2023 Aug 17;25(1):49. doi: 10.1186/s12968-023-00957-6. PMID 37587516
- [Derived] Bernhard B, Schnyder A, Garachemani D, Fischer K, Tanner G, Safarkhanlo Y, Stark AW, Schutze J, Pavlicek-Bahlo M, Greulich S, Johner C, Wahl A, Benz DC, Kwong RY, Grani C. Prognostic Value of Right Ventricular Function in Patients With Suspected Myocarditis Undergoing Cardiac Magnetic Resonance. JACC Cardiovasc Imaging. 2023 Jan;16(1):28-41. doi: 10.1016/j.jcmg.2022.08.011. Epub 2022 Oct 19. PMID 36599567
- [Derived] Fischer K, Obrist SJ, Erne SA, Stark AW, Marggraf M, Kaneko K, Guensch DP, Huber AT, Greulich S, Aghayev A, Steigner M, Blankstein R, Kwong RY, Grani C. Feature Tracking Myocardial Strain Incrementally Improves Prognostication in Myocarditis Beyond Traditional CMR Imaging Features. JACC Cardiovasc Imaging. 2020 Sep;13(9):1891-1901. doi: 10.1016/j.jcmg.2020.04.025. Epub 2020 Jul 15. PMID 32682718
- [Derived] Grani C, Eichhorn C, Biere L, Kaneko K, Murthy VL, Agarwal V, Aghayev A, Steigner M, Blankstein R, Jerosch-Herold M, Kwong RY. Comparison of myocardial fibrosis quantification methods by cardiovascular magnetic resonance imaging for risk stratification of patients with suspected myocarditis. J Cardiovasc Magn Reson. 2019 Feb 28;21(1):14. doi: 10.1186/s12968-019-0520-0. PMID 30813942